CLINICAL TRIAL: NCT04097561
Title: A Phase 1 Evaluation of the Safety of Belimumab in People With Idiopathic CD4 Lymphopenia and Autoantibodies (Phoebe)
Brief Title: Safety of Belimumab in People With Idiopathic CD4 Lymphopenia and Autoantibodies (Phoebe)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 190140; 19-I-0140
Record Dates: First submitted 2019-09-19; First posted 2019-09-20 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-03-27

CONDITIONS: Idiopathic CD4 Lymphopenia
Keywords: CD8 Counts; B-Cell Activating Factor (BAFF); Heterogeneous Disorder; Autoimmune Disease
MeSH Terms: conditions — T-Lymphocytopenia, Idiopathic CD4-Positive; Autoimmune Diseases | interventions — belimumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single arm, open-label (Experimental): Belimumab 10 mg/kg once every 2 weeks for 3 doses, and then once every 4 weeks for 5 doses, delivered via 1-hour intravenous (IV) infusion.
  Interventions: Biological: Belimumab

INTERVENTIONS:
Biological: Belimumab — Belimumab 10 mg/kg once every 2 weeks for 3 doses, and then once every 4 weeks for 5 doses, delivered via 1-hour intravenous (IV) infusion.

SUMMARY:
Background:

People with Idiopathic CD4 lymphopenia (ICL) have lower numbers of a type of white blood cell called CD4 cells. White blood cells fight against infections. Low levels of CD4 cells may make a person more likely to get sick. There are no approved treatments for ICL. Researchers think a drug called belimumab may be able to help in specific situations.

Objective:

To see if belimumab is safe for people with ICL.

Eligibility:

People ages 18-70 who have ICL and are participating in NIH protocol 09-I-0102 (EPIC)

Design:

Participants will be screened with:

Medical and medication history

Physical exam

Questionnaire about mental health and depression

Blood and urine tests

Participants will have a baseline visit. This will include some repeats of the screening tests. They may also have leukapheresis: Blood will be taken from a needle in one arm and passed through a machine that separates out the white blood cells. The rest of the blood will be returned through a needle in the other arm.

Participants will receive 8 doses of belimumab through IV: A needle will insert a thin plastic tube into an arm vein. Belimumab will be given through the IV line. The first 3 doses will be given every 2 weeks. The other 5 will be given once every 4 weeks. Participants will have a physical exam and blood and urine tests at each dosing visit. They will be monitored for up to 4 hours after the infusion.

Participants will have 3 follow-up visits, at around 8, 16, and 24 weeks after the last dose of belimumab. They will have a physical exam and blood and urine tests. Once they finish this protocol and they will continue to be followed under 09-I-0102 (EPIC study).

DETAILED DESCRIPTION:
Idiopathic CD4 lymphopenia (ICL) is characterized by persistent low CD4 counts, frequently in combination with CD8, natural killer, or B cell lymphopenia. It is considered a heterogeneous disorder with manifestations that can include autoimmunity, invasive fungal infections or infections with human papillomavirus, and malignancies typically related to infections. The exact etiology of ICL remains unclear and there is no specific treatment.

Recent data from our group revealed a high prevalence of antilymphocyte antibodies in many of the ICL patients evaluated. The targets of these antibodies remain unknown and are being investigated. On some occasions, these antibodies have the ability to cause antibody-dependent cytotoxicity or complement activation, both mechanisms that can cause cell death. Although it is unclear if these antibodies are the cause (or perhaps more likely the effect) of lymphopenia, it is plausible they play a significant pathogenic role and at a minimum may be hampering lymphocyte compensatory mechanisms for expansion and improved survival.

The immune deficiency and the unclear role of autoantibodies preclude aggressive immunosuppressive treatment (eg, corticosteroids) for ICL. Therefore, a rational approach to treatment is belimumab, a monoclonal antibody that targets Blys (also call BAFF for B-cell activating factor), expressed on activated B cells and plasma cells. Belimumab is approved by the United States Food and Drug Administration (FDA) for patients with systemic lupus erythematosus (SLE) who have evidence of autoantibodies and has shown efficacy in both reducing symptoms and leading to a modest decrease in autoantibodies.

In this open-label prospective single-arm study, ICL patients with laboratory evidence of antilymphocyte antibodies will be recruited. Belimumab will be administered by intravenous infusion for 6 months with an extended follow-up of an additional 6 months. Administration of the study drug will follow the SLE scheme of 10 mg/kg at study entry, 2 weeks, 4 weeks, and monthly thereafter (8 doses total). Three additional visits approximately every 2 months will complete the 52-week study. Clinical safety evaluations with immunologic and serologic testing will be performed at all study visits.

This protocol will assess the safety of belimumab in ICL and also help in better understanding the role of autoantibodies in ICL pathogenesis. This knowledge could substantially improve rationale and design of novel therapeutic interventions in ICL.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals must meet all of the following criteria to be eligible for study participation:

* Aged 18-70 years.
* Enrolled in study 09-I-0102.
* Has a documented diagnosis of ICL, defined as the following:

  * CD4 count < 300 cells/microliter in at least 2 separate measurements 6 weeks apart at any point in the past, AND
  * CD4 count < 300 cells/microliter within previous 90 days.
* Evidence for autoantibody positivity (eg, ANA or in the research flow method looking for antilymphocyte antibodies).
* Female participants of childbearing potential must agree to use adequate contraception when engaging in sexual activities that can result in pregnancy, beginning at day 0 (or day 30 for hormonal contraception) until 4 months after the last dose of belimumab.

Acceptable methods of contraception include the following:

* Hormonal contraception.
* Male or female condom.
* Diaphragm or cervical cap with a spermicide.
* Intrauterine device.

  * Able to provide informed consent.
  * Willing to allow samples to be stored for future research.

EXCLUSION CRITERIA:

Individuals meeting any of the following criteria will be excluded from study participation:

* Prior receipt of belimumab for any reason.
* Allergy to any component of belimumab formulation.
* HIV infection or other recognized congenital or acquired immunodeficiency.
* Current moderate or severe acute illness (eg, febrile illness, seizure, myocardial infarction, cerebrovascular accident, pulmonary embolism) or progressive serious infection related to ICL that, in the opinion of the principal investigator, would make the participant unsuitable for the study. Pre-existing infections that have been stable both clinically and with laboratory (eg, cryptococcal antigen titer or histoplasma antigen level) and radiographic evaluations on maintenance therapy over at least a year will be eligible.
* Untreated hepatitis B or C (acute or chronic).
* Active tuberculosis infection.
* Serum creatinine > 1.5 times the upper limit of normal (ULN).
* Hemoglobin < 8 g/dL.
* Alanine transaminase or aspartate transaminase > 2 times ULN.
* Serum IgG < 400 mg/L.
* Current use of systemic glucocorticosteroids, with the exception of corticosteroid nasal spray or inhaler and topical steroids.
* Any cancer diagnosis or autoimmune condition requiring systemic chemotherapy or immunomodulant-affecting antibody responses (eg, rituximab, ibrutinib), IV or SC Ig supplementation, radiation therapy, or any such treatment within the previous 6 months. Apremilast, Plaquenil, or nonsteroidal anti-inflammatory drugs will not be exclusionary.
* Severe depression. Psychiatry may be consulted prior to final eligibility decision.
* Infections (recently acquired or exacerbation of a chronic infection) that required new medications for management within the past 60 days.
* Receipt of any vaccination within the past 30 days.
* Pregnant.
* Breastfeeding.
* Any behavioral or substance use issue that would compromise appropriate follow up and participation in this study.

Concomitant diagnosis of SLE will not be exclusionary. Although SLE can be associated with lymphopenia, patients with lupus and extreme lymphopenia in the absence of cytotoxic or immunosuppressive medications and history of unusual infections will be eligible if they are participants of study 09-I-0102.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01-13 (Actual); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-03-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) that are possibly, probably, or definitely related to belimumab. | Week 2 through Week 48
  Incidence of AEs that are possibly, probably, or definitely related to belimumab.

SECONDARY OUTCOMES:
Evaluation of CD4 and CD8 counts at all study visits. | All study visits
  Evaluation of CD4 and CD8 counts at all study visits.
Evaluation of natural killer (NK) and B-cell counts at all study visits. | All study visits
  Evaluation of NK and B-cell counts at all study visits.
Evaluation of serum levels of BAFF at all study visits. | All study visits
  Evaluation of serum levels of BAFF at all study visits.
Evaluation of any known clinical autoimmune disease (eg, hemolytic anemia) or positive autoantibodies such as ANA at all study time points. | All study visits
  Evaluation of any known clinical autoimmune disease (eg, hemolytic anemia) or positive autoantibodies such as ANA at all study time points.

CONTACTS AND LOCATIONS:
Overall Officials: Irini Sereti, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2019-I-0140.html